CLINICAL TRIAL: NCT04161378
Title: Impact of Cardiac Rehabilitation Programs on Left Ventricular Remodeling After Acute Myocardial Infarction - the REHAB Trial
Status: Completed | Type: Observational
Sponsor: Cardio Med Medical Center (Industry)
Collaborators: George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures (Other); University Hospital of Targu Mures, Romania (Other)
Responsible Party: Sponsor
Other Study IDs: CM0121-REHAB
Record Dates: First submitted 2019-10-28; First posted 2019-11-13 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2019-11

CONDITIONS: Acute Myocardial Infarction; Non-ST Elevation Myocardial Infarction; Systemic Inflammation; Ventricular Remodeling; Acute Coronary Syndrome
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Ventricular Remodeling; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of venous blood samples at baseline and at 7 days after AMI for assessment of complete blood count, biochemistry, serum levels of hs-CRP, MMPs, IL6, NT-pro-BNP.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RHB-SG 01: Patients with early mobilization (< 2 days after the onset of symptoms)
  Interventions: Diagnostic Test: Cardiac imaging; Diagnostic Test: Laboratory analysis
- RHB-SG 02: Patients with delayed mobilization after AMI (>2 days after the onset of symptoms)
  Interventions: Diagnostic Test: Cardiac imaging; Diagnostic Test: Laboratory analysis

INTERVENTIONS:
Diagnostic Test: Cardiac imaging — * Transthoracic echocardiography
  * Late gadolinium enhancement CMR
Diagnostic Test: Laboratory analysis — * complete blood count
  * biochemistry
  * hs-CRP, MMPs, IL6, NT-pro-BNP

SUMMARY:
The aim of REHAB trial is to investigate the impact of early mobilization after AMI in reducing left ventricular remodeling, as assessed by cardiac magnetic resonance imaging. At the same time, the study aims to demonstrate the contribution of early mobilization to reduction of: systemic inflammation in the immediate post infarction phase, complication rates and mortality, in patients who had suffered a recent AMI, for a 1 year follow-up period.

DETAILED DESCRIPTION:
While the role of early mobilization in the immediate postinfarction period has been well demonstrated, little is known in present about the link between early mobilization and reduction of systemic inflammation. At the same time, the impact of early mobilization on regression of left ventricular remodeling has not been elucidated so far.

The study will be a single-center, observational, non-randomized study, which will be carried out in the Center of Advanced Research in Multimodal Cardiac Imaging Cardiomed, including 100 patients with AMI, presenting with either ST-segment elevation acute myocardial infarction (STEMI) or non-ST-segment elevation AMI (NSTEMI). According to the moment of mobilization after AMI patients will be distributed in two groups: group 1 - patients with early mobilization (<2 days after the onset of symptoms), and group 2 - subjects with delayed mobilization after AMI (>2 days after the onset of symptoms).

Each patient will be evaluated in terms of systemic inflammatory status in the immediate postinfarction phase, at baseline and at 7 days after AMI. In order to assess ventricular function and remodeling, extent of myocardial scar and transmurality index, late gadolinium enhancement CMR will be performed for each patient.

The study will be conducted over a period of 2 years, in which patients will be examined at baseline, and will be followed-up for 1 year for occurrence of MACE.

All patients will sign an informed written consent prior to study enrollment.

Study objectives:

Primary: to evaluate the impact of early mobilization after AMI on the ventricular remodeling in the post-infarction period, as assessed by CMR imaging. Secondary: to assess the rate of in-hospital mortality and the rate of repeated revascularization or MACE (including cardiovascular death or stroke) in patients with early mobilization as compared to those with delayed mobilization, and the effect of early mobilization on systemic inflammation in the immediate postinfarction phase.

Study Timeline:

* Baseline (day 0):
* Achieve written informed consent form all patients
* Check all inclusion/exclusion criteria
* Record demographic information, medical records, cardiovascular risk factors
* Perform and record physical examination and 12-lead ECG
* Laboratory analysis (CBC, routine biochemistry, inflammatory biomarkers, acute adhesion molecules)
* Transthoracic echocardiography / speckle tracking
* Visit 1 (day 7 / discharge from the hospital):
* hs-CRP assessment
* Visit 2 (month 1):
* LGE-CMR (myocardial fibrosis/scar, infarct size, transmurality, remodeling)
* Visit 3,4,5 (month 3,6,9):
* Record results of physical exam, medical records, ECG
* Transthoracic echocardiography / speckle tracking
* Final study visit (month 12):
* Record results of physical exam, medical records, ECG
* Transthoracic echocardiography / speckle tracking
* End-point assessment

Study procedures:

* Medical records, physical exam;
* Laboratory analysis (complete blood count, biochemistry, serum levels of hs-CRP, MMPs, IL6, NT-pro-BNP);
* Electrocardiography
* Transthoracic echocardiography for assessment of left ventricular systolic and diastolic performance, speckle tracking echocardiography, Dobutamine viability test
* Late gadolinium enhancement CMR for evaluation of ventricular function and remodeling, extent of myocardial scar and transmurality index.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AMI in the last 12 hours;
* Successful revascularization of the culprit artery within the first 12 hours after the onset of symptoms in STEMI or within first 48 hours in NSTEMI (according to the risk class);
* Signed written informed consent.

Exclusion Criteria:

* Patient refusal;
* Any condition that would contraindicate CMR examination;
* Women during pregnancy or lactation period;
* Women able to procreate without any contraceptive usage;
* Chronic kidney disease (glomerular filtration rate <60ml/min/1.73m2) or acute renal injury that requires hemodialysis;
* Any type of neoplasia documented in the last 3 years before randomization;
* Expectation of life < 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients with AMI, presenting with either ST-segment elevation acute myocardial infarction (STEMI) or non-ST-segment elevation AMI (NSTEMI).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Ventricular remodeling in the post-infarction period | Month 1
  LGE-CMR evaluation for myocardial fibrosis/scar, infarct size, transmurality, remodeling assessment.

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 12 months
  Rate of MACE at follow-up
Systemic inflammation in the immediate postinfarction phase | Day 7
  Inflammatory status evaluation via hs-CRP assessment at baseline and at 7 days from the acute event.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardio Med Medical Center, Târgu Mureş, Romania